CLINICAL TRIAL: NCT05167500
Title: Retrospective, Observational Study On The Efficacy And Safety Of Lorlatinib In ALK or ROS1 Metastatic Non-Small Cell Lung Cancer Patients Treated Within The Compassionate Use Program In Spain
Brief Title: Efficacy & Safety Study of Lorlatinib in ALK/ROS1 Metastatic NSCLC Patients With Compassionate Use Treatment
Acronym: LORLAPULM
Status: Completed | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 21/04_LORLAPULM
Record Dates: First submitted 2021-11-09; First posted 2021-12-22 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: Lung Diseases; Non small cell lung cancer; Metastatic disease; Lorlatinib; ALK alteration; ROS1 alteration
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Diseases; Neoplasm Metastasis | interventions — lorlatinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental : Lorlatinib inn ALK Or ROS1 Metastatic NSCLC patient: Patients with metastatic non-small cell lung cancer treated with lorlatinib who were included in the compassionate use program in Spain between November 2016 and February 2019 for those with an ALK alteration, and between November 2016 to March 2021 for those with ROS1 alteration.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — No treatment will be administered to the patient as an active treatment of this study. Only retrospective data about the patients treated in the compassion use program of Lorlatinib will be collected. The information below is related to Lorlatinib, target drug for the collection of data.
  Lorviqua 25 mg film-coated tablets.The recommended dose is 100 mg lorlatinib taken orally once daily. Treatment with lorlatinib is recommended as long as the patient is deriving clinical benefit from therapy without unacceptable toxicity. Dosing interruption or dose reduction may be required based on individual safety and tolerability.Lorlatinib should be permanently discontinued if the patient is unable to tolerate the 50 mg dose taken orally once daily.
  Other Names: Lorviqua

SUMMARY:
This is an observational, non-interventional, retrospective, multicentre and nationwide study. The information will be obtained retrospectively, in most cases when the treatment has already ended.

The primary objective of this study is determine the activity of lorlatinib (percentage of responses, duration of response, progression-free survival and time to treatment failure) of patients included in the compassionate use program in Spain.

DETAILED DESCRIPTION:
This is an observational, non-interventional, retrospective, multicentre and nationwide study. The information will be obtained retrospectively, in most cases when the treatment has already ended. In cases where the patient continues on the treatment, the researcher will not modify the clinical management of the patient by participating in the study.

Patients with metastatic non-small cell lung cancer treated with lorlatinib who were included in the compassionate use program in Spain between November 2016 and February 2019 for those with an ALK alteration, and between November 2016 to March 2021 for those with ROS1 alteration. According to the records of the Spanish centres participating in this program, approximately 145 patients have been included.

The primary objective of this study is determine the activity of lorlatinib (percentage of responses, duration of response, progression-free survival and time to treatment failure) of patients included in the compassionate use program in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic non-small cell lung cancer treated with lorlatinib who were included in the compassionate use program in Spain between November 2016 and February 2019 for those with an ALK alteration, and between November 2016 to March 2021 for those with ROS1 alteration.
* Patients must have been treated with at least one cycle of lorlatinib within the compassionate use program.
* Alive patients must have signed, dated the ethics committee approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.

Exclusion Criteria:

* Alive patients who refuse to sign and date an ethics committee approved written informed consent form.
* Patients who were accepted in the compassionate use program , but did not receive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic non-small cell lung cancer treated with lorlatinib who were included in the compassionate use program in Spain between November 2016 and February 2019 for those with an ALK alteration, and between November 2016 to March 2021 for those with ROS1 alteration. According to the records of the Spanish centres participating in this program, approximately 145 patients have been included.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of the first dose of lorlatinib treatment until the date of last follow up or death, assessed up to 60 months
  Progression-free survival defined as time from the first dose of lorlatinib to the first documentation of progression or death from any cause.
Duration of the response | From date of the first dose of lorlatinib treatment until the date of last follow up or death, assessed up to 60 months
  Duration of the response defined from the first documentation of tumor response to the first documentation of tumor progression or death from any cause.
Time to treatment failure | From date of the first dose of lorlatinib treatment until the date of last follow up or death, assessed up to 60 months
  Time to treatment failure defined as time from the first dose of lorlatinib to the moment of discontinuation of treatment for any cause, including tumor progression, toxicity or death

SECONDARY OUTCOMES:
Overall survival of ALK and ROS1 NSCLC patients | From date of the first dose of lorlatinib treatment until the date of last follow up or death, assessed up to 60 months
  Overall survival of ALK and ROS1 NSCLC patients from lorlatinib defined as time from the start of treatment until death or last follow-up
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From date of the first dose of lorlatinib treatment until the date of last follow up or death,assessed up to 60 months
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Calles, MD, Study Chair — Fundación GECP Investigator
Locations (25):
- Spain (25):
  - Hospital Clínico Santiago, Santiago de Compostela, A Coruña
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Centro Oncológico de Galicia, A Coruña, La Coruña
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital del Mar, Barcelona
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Universitario de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Fundación de Alcorcón, Madrid
  - Hospital Virgen del Rocio, Seville
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Universitari i Politécnic La Fe, Valencia
  - Hospital Clínico de Valencia, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundacion GECP studies — http://www.gecp.org